CLINICAL TRIAL: NCT06590103
Title: Effectiveness of Integrating Physically Active Learning Through Co-teaching in Extremadura: ACTIVA-MENTE Project
Acronym: ACTIVA-MENTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Collaborators: Consejería de Educación, Ciencia y Formación Profesional. Junta de Extremadura (Unknown)
Responsible Party: Principal Investigator, David Sanchez Oliva, Assistant Professor, University of Extremadura
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08/2024
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Physical Activity; Adolescents; Physical Fitness
Keywords: Physuca active learning; Motivational variables; Sedentary time; Academic indicators
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physically Active Lessons. (Experimental): Physically Active Learning: consists of incorporating physical activity (usually of moderate-vigorous intensity) into the educational content taught in non-physical education academic classes.
  Interventions: Behavioral: Physically Active Lessons
- Control group (No Intervention): The control group will receive the usual academic classes without any methodological modification during the intervention period.

INTERVENTIONS:
Behavioral: Physically Active Lessons — Physically active learning: this type of intervention is carried out once a week for 1 hour outside the classroom. The teachers of the corresponding subject (with the support of the Physical Education teacher) are in charge of designing and delivering the physically active classes.
  Arms: Physically Active Lessons.

SUMMARY:
Study based on a school-based physically active learning intervention during the school day on physical activity, fitness, health and education outcomes in adolescents.

DETAILED DESCRIPTION:
Activamente is a quasi-experimental study coordinated by fully qualified researchers in physical activity and sport sciences from the University of Extremadura (UEX), Spain. This study is aimed at students from 1st to 4th year of Secondary Education (11-16 years old), belonging to 10 schools in the Autonomous Community of Extremadura. Each school will have five experimental groups and five control groups. Thus, there will be 50 experimental groups (n=1100) and 50 control groups (n=1100). The intervention will last 8 months, and will consist of one component, which is the inclusion of one physically active class per week.

Before and after the intervention, physical activity and sedentary time will be assessed by activity bracelets, health-related fitness levels by field tests, body composition parameters by anthropometry, academic performance by school grades, positive health (quality of life and self-perception of health) by questionnaire, and cognitive parameters (executive functions) by specific cognition tests. In addition, two intermediate measures of physical activity levels and sedentary time will be measured.

At the end of the intervention the investigators will determine changes in the main outcome variables. Also, the main hypotheses raised will be:

1. Students belonging to the experimental group will improve physical activity and decrease sedentary time during the school day when compared to students belonging to the control group.
2. The students belonging to the experimental group will improve in the markers of physical and psychological health when compared to the students belonging to the control group.
3. Students in the experimental group will improve their academic and cognitive indicators when compared to students in the control group.
4. Students belonging to the experimental group will improve school climate and motivational variables in academic classes when compared to students belonging to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in 1st, 2nd, 3rd and 4th year of ESO.
* Adolescents with informed consent signed by the family/guardian.
* Schools with at least 210 students enrolled in 1st, 2nd, 3rd and 4th year of ESO.
* Schools belonging to the Autonomous Community of Extremadura.

Exclusion Criteria:

* Adolescents with any physical disability or health condition that may limit physical activity levels.
* Schools participating in any other physical activity or health promotion program.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Physical activity and sedentary time | 8 months
  Physical activity and sedentary time will be measured by the Fitbit activity wristband version 6.0.

SECONDARY OUTCOMES:
Cardiorespiratory capacity | 8 months
  The 20-metres shuttle run test will be used to assess cardiorespiratory fitness. Participants will run the 20-metre distance to the rhythm of a recording. The initial speed is 8.5 km/h and will be increased by 0.5 km/h per section. The race will end when the participant stops due to fatigue or when he/she fails to cross the marked lines to the rhythm of the acoustic signals on two consecutive occasions. The last stage or half stage completed by the competitor will be scored.
Musculoskeletal capacity of Upper body | 8 months
  The hand grip test will be used to assess musculoskeletal capacity of upper body. The test shall be performed twice with each hand alternately. The maximum score of each hand in kilograms shall be recorded and the mean value between them shall be calculated.
Musculoskeletal capacity of lower body | 8 months
  Standing broad jump shall be used to assess the musculoskeletal capacity of the lower limbs. The participant shall stand behind a line with feet shoulder width apart. The participant is then asked to jump forward as far as possible with both feet. If he/she rests his/her hands or lifts his/her feet off the ground when landing, the test is invalid. The test shall be performed twice, and the best score recorded in centimetres.
Body mass index | 8 months
  Weight and height will be combined to report BMI in kg/m^2.
Health status | 8 months
  General health status is assessed using the visual analog scale that includes the five-dimensional, three-level EuroQol questionnaire (EQ-5D-3L) (Ravens-Sieberer et al., 2010). For this, students are asked to assign a score from 0 to 100 to indicate their perception of their general health status.
School engagement | 8 months
  The engagement scale (UWES-S-9) will be used to evaluate school engagement. The UWES-S-9 is composed of nine items that reflect the three dimensions of engagement: (i) vigor; (ii) absorption; and (iii) dedication, each dimension is represented by three items that will be evaluated through a Likert-type scale, ranging from "never" (0 points) to "always" (6 points).
Learning perception | 8 months
  The perception of learning in the different subjects worked on will be evaluated by means of a questionnaire composed of eight items. Items 1- 4 will assess the dimension "perceived learning" and items 5-8 will measure the dimension "satisfaction with learning". All items will be scored according to a five-point Likert scale, where "1" is (strongly disagree) and "5" is (strongly agree).
Academic performance | 8 months
  Academic performance will be evaluated through the marks reported by the schools before and after the intervention.
Novelty | 8 months
  Novelty will be assessed through the Novelty Need Satisfaction Scale. Five of the 19 questions that make up the original scale will be selected and participants will be asked to answer them on a Likert-type scale where 1 = "strongly disagree" and 5 = "strongly agree".
School climate | 8 months
  School climate will be assessed using the students' perception of school climate scale (PACE-33). Fifteen items will be evaluated. All items will be scored according to a five-point Likert scale, where "1" is (strongly disagree) and "5" is (strongly agree).
Sociodemographic characteristics | 8 months
  Sociodemographic characteristics will be measured through the Spanish-adapted version III of The Family Affluence Scale. This scale is composed of six questions . Each question is scored on a categorical scale, and the sum of the scores from the six items result in an aggregate index ranging from 0 to 13.
Teachers' perceptions about the feasibility of the intervention program. | 8 months
  Perception about the suitability and the development of the intervention program (perceptions, barriers, points to improve, strengths...) a semi-structured interview will be conducted with the teachers involved in the intervention.
Students' perceptions about the feasibility of the intervention program. | 8 months
  A discussion group will be developed for each of the proposed interventions with a subsample of students, in order to obtain information on the suitability and development of the intervention programme (perceptions, barriers, areas for improvement, strengths, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Cáceres, Spain